CLINICAL TRIAL: NCT07222436
Title: Circulating Tumor DNA in High Risk Localized Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: The Beckwith Institute (Other)
Responsible Party: Principal Investigator, Leonard Appleman, Associate Professor of Medicine, University of Pittsburgh
Other Study IDs: HCC 25-054
Record Dates: First submitted 2025-10-27; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; ctDNA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating free DNA (cfDNA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, non-therapeutic translational biomarker study will collect blood in patients with high risk localized prostate cancer prior to prostatectomy.

DETAILED DESCRIPTION:
The Vogelstein lab has developed a highly sensitive, tumor-informed method of detecting circulating free DNA (cfDNA) shed by solid tumors. Plasma will be assayed for ctDNA using the SaferSeqS tumor-informed assay, employing DNA sequences derived from prostatectomy specimens. The abundance and molecular characteristics of ctDNA will be evaluated for a pilot group of 12-24 patients using an adaptive statistical design.

ELIGIBILITY:
Inclusion Criteria:

1. Must have histologically confirmed prostate cancer.
2. Age ≥ 18 years.
3. ECOG performance status of 0-1.
4. Must have the ability to understand and the willingness to sign a written informed consent document.
5. Willing to provide serial blood samples for the study.
6. Willing to provide tumor tissue (prostatectomy for primary cohort; prostatectomy or biopsy for exploratory cohort) for correlative studies which will compare ctDNA to tumor specimens.
7. Primary Cohort: High-risk localized prostate adenocarcinoma defined as one or more of the following:

   o Clinical stage ≥ cT3a, Grade Group 4 or 5 (Gleason sum 8-10), and PSA ≥ 20

   *Non-bulky pelvic lymphadenopathy and indeterminate findings on staging imaging (CT, bone scan, PSMA PET CT) are allowed if the surgeon believes RP is appropriate.
8. Exploratory Cohort: Men with a diagnosis of prostate adenocarcinoma and one of the following:

   * Localized prostate adenocarcinoma on active surveillance
   * Biochemically-recurrent prostate adenocarcinoma after definitive local therapy
   * Hormone-sensitive, metastatic prostate adenocarcinoma
   * Metastatic CRPC

Exclusion Criteria:

1. History of another primary cancer within the last 3 years, except for non-melanomatous skin cancer.
2. Receiving androgen deprivation or other systemic therapy for prostate cancer.
3. Medical condition or social situation that may preclude adherence to the protocol.

   -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high risk localized prostate cancer prior to prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
ctDNA detection | Up to 2 years
  Detection of ctDNA by assay in blood collected prior to radical prostatectomy using the Vogelstein lab assay. This assay is a highly sensitive, tumor-informed method of detecting circulating free DNA (cfDNA) shed by solid tumors that has shown prognostic value for recurrence and predictive for benefit of adjuvant chemotherapy.

SECONDARY OUTCOMES:
ctDNA abundance | Up to 2 years
  Quantification of ctDNA by assay in blood collected prior to radical prostatectomy using the Vogelstein lab assay. This assay is a highly sensitive, tumor-informed method of detecting circulating free DNA (cfDNA) shed by solid tumors that has shown prognostic value for recurrence and predictive for benefit of adjuvant chemotherapy.
serum PSA recurrence | At 6 weeks post-operative
  The detection of prostate-specific antigen (PSA) levels that rise after initial treatment for prostate cancer. This can indicate a regrowth of cancer cells or a biochemical recurrence, meaning that while the cancer may not be visible on imaging, it is still present in the body.
serum PSA recurrence | At 6 months post-operative
  The detection of prostate-specific antigen (PSA) levels that rise after initial treatment for prostate cancer. This can indicate a regrowth of cancer cells or a biochemical recurrence, meaning that while the cancer may not be visible on imaging, it is still present in the body.
serum PSA recurrence | At 12 months post-operative
  The detection of prostate-specific antigen (PSA) levels that rise after initial treatment for prostate cancer. This can indicate a regrowth of cancer cells or a biochemical recurrence, meaning that while the cancer may not be visible on imaging, it is still present in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No